CLINICAL TRIAL: NCT00552903
Title: Randomised Trial of Health Coaching in Secondary Prevention of Diabetes and Heart Disease
Acronym: TerVa
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Paijat-Hame Hospital District (Other)
Collaborators: Sitra, the Finnish Innovation Fund (Other); Pfizer (Industry); Tampere University (Other)
Responsible Party: Dr Martti Talja, Päijät-Häme Health and Welfare Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHKS-Z80
Record Dates: First submitted 2007-11-01; First posted 2007-11-02 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure; Coronary Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure; Coronary Disease | interventions — Counseling

ARMS (2):
- 1 (Experimental): Active intervention - personal health coaching provided
  Interventions: Behavioral: Health coaching
- 2 (No Intervention): Control arm - no intervention, data on health outcomes collected at baseline (entry to the study) and during the 12 month follow-up

INTERVENTIONS:
Behavioral: Health coaching — Personal health coach providing advice and counselling by telephone, weekly contacts
  Other Names: Counseling, health education
  Arms: 1

SUMMARY:
A randomised trial with individual patients as units of observation will be carried out. Health coaching is used to modify health behaviour and thus improve disease control and health status, as well as use of health care services. A personal health coach is assigned to each patient and they are in weekly contact through telephone. The intervention lasts for 12 months. No intervention is offered to the patients in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes (medication and HbA1c>7% and no cardiovascular disease), coronary artery disease (history of myocardial infarction or revascularisation) or heart failure (NYHA II-III and admitted in a hospital for the condition within 2 years)
* Aged 45 years or older
* Resident in the Päijät-Häme health care district

Exclusion Criteria:

* Classified as ineligible by primary care physician
* Unable to co-operate or participate in health coaching
* Major elective surgery planned within 6 months
* History of major surgery within past 2 years
* Life expectancy <1 year
* Pregnancy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Blood pressure at target level (140/85 or lower), total cholesterol at target level (4.5 mmol/l or lower), LDL cholesterol at target level (2.5 mmol/l or below), waist circumference at target level (<=94 men, <=80 cm women) | 12 months from start of intervention
For patients with diabetes: blood HbA1c at target level (7% or less) | 12 months from start of intervention

SECONDARY OUTCOMES:
Improvement in body mass index, health-related quality of life (15D instrument), amount of exercise, diet, smoking cessation; for patients with heart failure also use of emergency services and NYHA class | 12 months from start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martti Talja, MD, Principal Investigator — Päijät Häme Central Hospital; Ilmo Parvinen, MD, Study Chair — Sitra, the Finnish Innovation Fund
Locations (1):
- Päijät-Hämeen Sosiaali - ja Terveysyhtymä, Lahti, Finland

REFERENCES:
- [Derived] Mustonen E, Horhammer I, Patja K, Absetz P, Lammintakanen J, Talja M, Kuronen R, Linna M. Eight-year post-trial follow-up of morbidity and mortality of telephone health coaching. BMC Health Serv Res. 2021 Nov 15;21(1):1237. doi: 10.1186/s12913-021-07263-w. PMID 34781936
- [Derived] Mustonen E, Horhammer I, Absetz P, Patja K, Lammintakanen J, Talja M, Kuronen R, Linna M. Eight-year post-trial follow-up of health care and long-term care costs of tele-based health coaching. Health Serv Res. 2020 Apr;55(2):211-217. doi: 10.1111/1475-6773.13251. Epub 2019 Dec 29. PMID 31884682
- [Derived] Oksman E, Linna M, Horhammer I, Lammintakanen J, Talja M. Cost-effectiveness analysis for a tele-based health coaching program for chronic disease in primary care. BMC Health Serv Res. 2017 Feb 15;17(1):138. doi: 10.1186/s12913-017-2088-4. PMID 28202032
- [Derived] Patja K, Absetz P, Auvinen A, Tokola K, Kyto J, Oksman E, Kuronen R, Ovaska T, Harno K, Nenonen M, Wiklund T, Kettunen R, Talja M. Health coaching by telephony to support self-care in chronic diseases: clinical outcomes from The TERVA randomized controlled trial. BMC Health Serv Res. 2012 Jun 10;12:147. doi: 10.1186/1472-6963-12-147. PMID 22682298